CLINICAL TRIAL: NCT02389348
Title: A Proof-of-concept Study to Assess the Effect of a Range of Doses of Combined Therapy With OZ439 and DSM265 Against Early Plasmodium Falciparum Blood Stage Infection in Healthy Participants
Brief Title: A Phase Ib Induced Malaria Infection Study With the Combination of OZ439 and DSM265
Acronym: OZ/DSMCombo
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Q-Pharm Pty Limited (Industry); QIMR Berghofer Medical Research Institute (Other); Clinical Network Services (CNS) Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QP14C12
Record Dates: First submitted 2015-02-20; First posted 2015-03-17 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Malaria
Keywords: Induced blood stage malaria
MeSH Terms: conditions — Malaria | interventions — DSM265

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- combination OZ439 and DSM265 (Experimental): Subjects will receive 1800 P falciparum infected red blood cells. Development of parasitemia will be monitored by quantitative PCR. When the parasitemia reached the threshold of 1000 p/ml subjects will receive a single oral dose of OZ439 and DSM265.
  Subsequent doses in subsequent cohort(s) will be determined following a review of observed OZ439 and DSM265 safety, and pharmacokinetic and pharmacodynamic interaction outcomes as well as the activity of the drugs as defined by parasite clearance kinetics.
  Interventions: Drug: DSM265; Drug: OZ439

INTERVENTIONS:
Drug: DSM265 — Single oral doses of DSM265
Drug: OZ439 — Single oral doses of OZ439

SUMMARY:
This is a single-centre, open-label, dose finding study using induced blood stage malaria (IBSM) infection to characterize the pharmacodynamic interaction between OZ439 and DSM265, administered around 120 minutes apart for treatment of early Plasmodium falciparum blood stage infection. The study will be conducted in up to three cohorts (n=8 per cohort) using different doses of OZ439 and DSM265. The doses of OZ439 and DSM265 that will be investigated in the first cohort will be 200 mg of OZ439 and 100mg of DSM265, both administered as single doses around 120 minutes apart. Subsequent doses in subsequent cohort(s) will be determined following a review of observed OZ439 and DSM265 safety, and pharmacokinetic and pharmacodynamic interaction outcomes, particularly the antimalarial activity of the drugs given in combination as defined by parasite clearance kinetics. The doses used in Cohort 2 and 3 may be adjusted but will not exceed the maximum acceptable doses predefined for this study (which are 400 mg for DSM265 and 500mg for OZ439) as determined in previous safety and pilot efficacy studies. The dose will be determined by the funding sponsor and the principal investigator (PI) following Safety Review team (SRT) and scientific evaluation. If no safe alternative dose can be determined the option exists to curtail the study to less than three cohorts.

Each participant in the cohort will be inoculated on Day 0 with ~1,800 viable parasites of Plasmodium falciparum-infected human erythrocytes (BSPC) administered intravenously. On an outpatient basis, participants will be monitored daily via phone call and then daily (AM) from day 4 (until PCR positive for presence of malaria parasites). Once PCR positive they will be monitored twice-daily morning (AM) and evening (PM) until treatment, for adverse events and the unexpected early onset of symptoms, signs or parasitological evidence of malaria. On the day designated for commencement of treatment, as determined by qPCR results, participants will be admitted to the study unit and monitored. The threshold for commencement of treatment will be when PCR quantification of all participants is = 1,000 parasites/mL. If the PCR quantification of any participant is = 5,000 parasites/mL and is accompanied by a clinical symptom score >5, or if clinical or parasitological evidence of malaria occurs in any participant before all participants have reached the treatment threshold (PCR quantification of = 1,000), then treatment of that participant will begin within a 24 h period.

Following treatment with OZ439 and DSM265, participants will be followed up as inpatients for at least 48 hours to ensure tolerance of the treatment and clinical response, then if clinically well on an outpatient basis for safety and clearance of malaria parasites via PCR.

Compulsory commencement of treatment with Riamet® (artemether-lumefantrine) will occur on study day 16 ±3 days post OZ439 and DSM265 treatment unless required earlier. Early standard anti-malarial drug intervention can occur if either poor responses or fast responses are seen following OZ439 and DSM265 treatment. This is to ensure participant safety and to avoid participant inconvenience if useful data cannot be obtained. A poor response is defined as a decrease in parasitaemia of less than 20% from baseline by 3 days post OZ439 and DSM265 treatment. A fast response occurs when, within the seven day period following the treatment, two consecutive PCR assessments in 48 hours are negative. However, pre-emptive treatment with Riamet® can commence whenever deemed necessary by the investigator. Participants will be monitored, either in clinic, or by telephone for three days to ensure adherence to Riamet® therapy.

Participants will be treated with a single dose (45 mg) of primaquine as described in section 4.3 in this protocol at the end of their Riamet® treatment if gametocytes are identified, to ensure complete clearance of any gametocytes present.

Adverse events will be monitored via telephone monitoring, within the clinical research unit, and on outpatient review after malaria challenge inoculation and antimalarial study drugs administration. Blood samples for safety evaluation, malaria monitoring, and red blood cell antibodies will be drawn at screening and/ or baseline and at nominated times after malaria challenge.

ELIGIBILITY:
Inclusion Criteria:

Demography

* Adults (male and non-pregnant and non-lactating females) participants between 18 and 55 years of age, inclusive who do not live alone (from Day 0 until at least the end of the antimalarial drug treatment) and be contactable and available for the duration of the trial (maximum of 4 months).
* Female participants of childbearing potential must have adequate contraception in place (see section 6.7) for the duration of the study and extended duration, and have negative results on a serum or urine pregnancy test done before administration of study product. Males prepared to use adequate contraception for the duration of study and extended duration (See section 6.7)
* Body weight, minimum 50.0 kg, body mass index between 18.0 and 32.0 kg/m2, inclusive.

Health status

* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Normal vital signs after 5 minutes resting in supine position:

  * 95 mmHg < systolic blood pressure (SBP) <140 mmHg,
  * 50 mmHg < diastolic blood pressure (DBP) <90 mmHg,
  * 40 bpm< heart rate (HR) <100 bpm.
  * Oral body temperature between 35.0 - 37.5◦C
* Normal standard 12-lead electrocardiogram (ECG) after 5 minutes resting in supine position, QTcF=450 ms with absence of second or third degree atrioventricular block or abnormal T wave morphology.
* Laboratory parameters within the normal range, unless the Investigator considers an abnormality to be clinically irrelevant for healthy participants enrolled in this clinical investigation. More specifically for serum creatinine, hepatic transaminase enzymes (aspartate aminotransferase, alanine aminotransferase), and total bilirubin (unless the Participant has documented Gilbert syndrome) should not exceed the upper laboratory normal and haemoglobin must be equal or higher than the lower limit of the normal range, Regulations
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion Criteria:

Medical history and clinical status

* Any history of malaria or participation to a previous malaria challenge study
* Must not have travelled to or lived (>2 weeks) in a malaria-endemic country during the past 12 months or planned travel to a malaria-endemic country during the course of the study.
* Has evidence of increased cardiovascular disease risk (defined as >10%, 5 year risk) as determined by the method of Gaziano et al. (1). Risk factors include sex, age, systolic blood pressure (mm/Hg), smoking status, body mass index (BMI, kg/m2) and reported diabetes status.
* History of splenectomy.
* Presence or history of drug hypersensitivity, or allergic disease diagnosed and treated by a physician or history of a severe allergic reaction, anaphylaxis or convulsions following any vaccination or infusion. Lactose Intolerant.
* Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immunodeficiencies), insulin-dependent Type 1 and Type 2 and NIDDM diabetes (excluding glucose intolerance if Exclusion criteria 3 is met), progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, psoriasis, rheumatoid arthritis, uncontrolled asthma, epilepsy or obsessive compulsive disorder, skin carcinoma excluding non-spreadable skin cancers such as basal cell and squamous cell carcinoma.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study. The Investigator should make this determination in consideration of the subject's medical history and/or clinical or laboratory evidence of any of the following:

  * Inflammatory bowel disease, ulcers, gastrointestinal or rectal bleeding in the last 6 months;
  * Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
  * Pancreatic injury or pancreatitis in the last 6 months;
* Participants with history of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis. including depression or receiving psychiatric drugs or who has been hospitalized within the past 5 years prior to enrollment for psychiatric illness, history of suicide attempt or confinement for danger to self or others.
* Frequent headaches and/or migraine, recurrent nausea, and/or vomiting (more than twice a month).
* Presence of acute infectious disease or fever (e.g., sub-lingual temperature = 38.5°C) within the five QP14C12_OZ439-DSM265 MMV Challenge Protocol_v1.1_26Nov 2014 Page 9 of 71 days prior to inoculation with malaria parasites.
* Evidence of acute illness within the four weeks before trial prior to screening that the Investigator deems may compromise subject safety.
* Significant inter-current disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urin analysis.
* Participant has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion, e.g. gastrectomy, diarrhoea.
* Participation in any investigational product study within the 12 weeks preceding the study.
* Participation in any research study involving to be desired blood sampling (more than 450 mL/ unit of blood), or blood donation to Australian Red Cross (or other) blood bank during the 8 weeks preceding the reference drug dose in the study.
* Participant unwilling to defer blood donations to the ARCBS for 6 months.
* Blood donation, any volume, within 1 month before inclusion.
* Medical requirement for intravenous immunoglobulin or blood transfusions.
* Participant who has ever received a blood transfusion.
* Symptomatic postural hypotension at screening, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure =20 mmHg within 2-3 minutes when changing from supine to standing position.
* History or presence of alcohol abuse (alcohol consumption more than 40 g per day, ( 3 standard drinks per day) or drug habituation, or any prior intravenous usage of an illicit substance.
* Smoking more than 5 cigarettes or equivalent per day and unable to stop smoking during the study.
* Ingestion of any poppy seeds within the 24 hours prior to the screening blood test (participants will be advised by phone not to consume any poppy seeds in this time period).
* Excessive consumption of beverages containing xanthine bases, including red bull, chocolate, etc, (eg, more than 400 mg of caffeine per day (more than 4 cups or glasses per day).

Interfering substance

* Any medication (including St John's Wort) within 14 days malaria inoculum (day 0) or within 5 times the elimination half-life (whichever is longer) of the medication.
* Any vaccination within the last 28 days.
* Any corticosteroids, anti-inflammatory drugs, immunomodulators or anticoagulants. Any participant currently receiving or having previously received immunosuppressive therapy, including systemic steroids including adrenocorticotrophic hormone (ACTH) or inhaled steroids in dosages which are associated with hypothalamic-pituitary-adrenal axis suppression such as 1 mg/kg/day of prednisone or its equivalent or chronic use of inhaled high potency corticosteroids (budesonide 800 µg per day or fluticasone 750 µg).
* Any recent or current systemic therapy with an antibiotic or drug with potential antimalarial activity (chloroquine, piperaquine, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, hydroxychloroquine, etc.).

General conditions

* Any participant who, in the judgment of the Investigator, is likely to be noncompliant during the study, QP14C12_OZ439-DSM265 MMV Challenge Protocol_v1.1_26Nov 2014 Page 10 of 71 or unable to cooperate because of a language problem or poor mental development.
* Any participant in the exclusion period of a previous study according to applicable regulations.
* Any participant who lives alone (from Day 0 until at least the end of the antimalarial drug treatment).
* Any participant who cannot be contacted in case of emergency for the duration of the trial and up to 2 weeks following end of study visit.
* Any participant who is the Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
* Any participant without a good peripheral venous access. Biological status
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, antihepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab),
* Participant is found to be G6PD deficient
* Any drug listed in Table 2 in the urine drug screen unless there is an explanation acceptable to the medical investigator (e.g., the participant has stated in advance that they consumed a prescription or OTC product which contained the detected drug) and/or the Participant has a negative urine drug screen on retest by the pathology laboratory.
* Positive alcohol urine or breath test. Specific to the study
* Cardiac/QT risk:

  * Known pre-existing prolongation of the QTcB interval considered clinically significant,
  * Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc-interval or any clinical condition known to prolong the QTc interval. History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia. Electrolyte disturbances,particularly hypokalaemia, hypocalcaemia or hypomagnesaemia,
  * Electrocardiogram (ECG) abnormalities in the standard 12-lead ECG (at screening) which in the opinion of the Investigator is clinically relevant or will interfere with the ECG analysis,
  * A history of clinically significant ECG abnormalities.
* Known hypersensitivity to OZ439 or DSM265 or any of its excipients or excipients or artemether or other artemisinin derivatives, lumefantrine, or other arylamino alcohols.
* Unwillingness to abstain from consumption of citrus (grapefruit, Seville orange, etc.) as well as quinine containing foods/beverages such as tonic water, lemon bitter, from inoculation (Day 0) to the end of the malaria treatment or as advised by the clinical personnel.
* Use of any prescription drugs, herbal supplements, within four (4) weeks prior to initial dosing, and/or over-the-counter (OTC) medication, dietary supplements (vitamins included) within two (2) weeks prior to initial dosing (note that diazepam interferes with the analysis of DSM265 and should not have been used for 8 weeks prior to initial dosing). If needed, (i.e. an incidental and limited need) paracetamol is acceptable up 4 g/day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
PK/PD relationship on clearance of P falciparum parasites from the blood | From treatment administration to clearance of parasites or administration of Standard of Care therapy, whichever comes first, and up to 42 days following inoculum
  The Parasite Reduction Ratio (PRR) is estimated using the slope of the optimal fit of the log-linear relationship of the parasitemia decay.

SECONDARY OUTCOMES:
Incidence, relation to study drug and severity of AE | From challenge inoculum and up to 42 days following inoculum
  Assessment of tolerability and safety of OZ439 and DSM265 in the challenge model
Cmax, Tmax, AUC of DSM265 and OZ439 | From Drug administration up to 42 days following inoculum
  Appropriate PK parameters will be determined including non-compartmental and modeling characterisation

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, Prof, Principal Investigator — Q-Pharm Pty Limited
Locations (1):
- Q-Pharm Clinics, Herston, Queensland, Australia

REFERENCES:
- [Derived] Dini S, Zaloumis SG, Price DJ, Gobeau N, Kummel A, Cherkaoui M, Moehrle JJ, McCarthy JS, Simpson JA. Seeking an optimal dosing regimen for OZ439/DSM265 combination therapy for treating uncomplicated falciparum malaria. J Antimicrob Chemother. 2021 Aug 12;76(9):2325-2334. doi: 10.1093/jac/dkab181. PMID 34179977
- [Derived] McCarthy JS, Ruckle T, Elliott SL, Ballard E, Collins KA, Marquart L, Griffin P, Chalon S, Mohrle JJ. A Single-Dose Combination Study with the Experimental Antimalarials Artefenomel and DSM265 To Determine Safety and Antimalarial Activity against Blood-Stage Plasmodium falciparum in Healthy Volunteers. Antimicrob Agents Chemother. 2019 Dec 20;64(1):e01371-19. doi: 10.1128/AAC.01371-19. Print 2019 Dec 20. PMID 31685476